CLINICAL TRIAL: NCT02581969
Title: Extension at 10 Years of the: "Observational Study Evaluating Efficacy and Costs of Secondary Prophylaxis vs On-demand Therapy With Kogenate Bayer in Patients With Severe Haemophilia A." POTTER-10
Brief Title: Extension at 10 Years of the: "Observational Study Evaluating Efficacy and Costs of Secondary Prophylaxis vs On-demand Therapy With Kogenate Bayer in Patients With Severe Haemophilia A."
Acronym: POTTER 10
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18251
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Hemophilia A
Keywords: Hemophilia A, Congenital
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prophylaxis: Prophylaxis group: treatment is based on regularly repeated infusions of clotting factor, 20-30 IU/kg -3 times a week
  Interventions: Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- On-demand: On-demand group: treatment administered when bleeding episode occur
  Interventions: Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Administered 20-30 IU/kg 3 times a week
  Groups: Prophylaxis
Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Administered only for bleeding episodes
  Groups: On-demand

SUMMARY:
Following the performance of the POTTER observational study, whose primary objective was to collect data on the benefits of secondary prophylaxis versus on demand treatment in terms of prevention of bleeding episodes, the present study aims to extend the observation time up to 10 years, of the same population involved in the previous study.

The present study has been designed to allow a focus on long term disease-related damage at joint level in subjects with severe haemophilia A, as well as on the pharmacoeconomics impact of the two different treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Completion of follow-up in the original Potter study without having being excluded from the Intention To Treat efficacy analysis of the primary endpoint;
* Written informed consent specifically issued for the 5-year extension.

Exclusion Criteria:

* Switching of treatment to a Factor VIII concentrate different from Kogenate Bayer/Helixate NexGen after the end of the previous follow-up period.

Ages: 17 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of approximately 50 patients with a diagnosis of severe haemophilia A (FVIII < 1%) , who are already on Kogenate Bayer treatment ongoing for long-term secondary prophylaxis or on-demand therapy and have properly completed the follow-up in the original Potter study are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Number of joint bleeding episodes per year | 5 years period

SECONDARY OUTCOMES:
Total number of bleeding episodes per year | 5 years period
Total amount of Recombinant Factor VIII consumption | 5 years period
Changes of prophylaxis dose | 5 years period
Changes of frequency of infusions | 5 years period
Musculoskeletal evaluation by calculating the World Federation of Haemophilia Orthopedic Joint Score (Gilbert score) | 5 years period
Proportions of patients who will change the therapeutic regimen during the study | 5 years period
Musculoskeletal evaluation by calculating the Radiological score (Pettersson Score) | 5 years period
Evaluating the Questionnaires of Health-Related Quality of Life _Haemo Quality of Life (HaemoQol) | 5 years period
Evaluating the Questionnaires of Health-Related Quality of Life _Short Form 36 questions (SF36) | 5 years period
Evaluating the Questionnaires of Health-Related Quality of Life _ Euro Quality 5 Dimension (EQ5D) | 5 years period
Number of days missed from work or school of patients and caregivers because of all the events haemophilia-related | 5 years period
Number of patients with poor compliance | 5 years period
Number of patients with adverse events | 5 years period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Italy